CLINICAL TRIAL: NCT07050953
Title: Prevalence of Ascending Aortic Dilation in Sports Medicine
Acronym: PRAADS
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: Ao-TTE
Record Dates: First submitted 2025-03-21; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-03

CONDITIONS: Aortic Aneurysm; Athlete
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Recreational and competitive Athletes: All athletes aged over 10 years consulting for routine sports medicine evaluation, regardless of sport type or performance level.
  Interventions: Other: focused cardiac ultrasound

INTERVENTIONS:
Other: focused cardiac ultrasound — A focused cardiac ultrasound will be performed to measure the dimensions of ascending aorta

SUMMARY:
This study aims to assess the prevalence of ascending aortic dilation in athletes from the general population undergoing routine sports medicine evaluation. It also evaluates the predictive factors and the reproducibility of focused cardiac ultrasound.

DETAILED DESCRIPTION:
Ascending aortic dilation is a potentially serious and underdiagnosed cardiovascular condition, particularly in the context of physical activity. While its prevalence has been studied in elite athletes, little data is available regarding the general athletic population undergoing routine sports medicine evaluation. This study aims to investigate the prevalence of ascending aortic dilation in a general population of recreational and competitive athletes.

This is an observational study conducted at the Sports Medicine Department of Caen University Hospital (France). The study will include athletes over the age of 10 who consult for a pre-participation medical evaluation. A focused cardiac ultrasound (FCU) protocol targeting the ascending aorta will be systematically performed using a portable ultrasound device during routine clinical assessment. When indicated, a standard transthoracic echocardiography (TTE) will be used as the reference method for comparison.

The primary objective of the study is to estimate the prevalence of ascending aortic dilation in this population. The secondary objective is to explore potential predictive factors, including cardiovascular risk factors and exercise history.

This study may help clarify the utility of FCU as a screening tool in sports medicine and contribute to improved early detection of aortic abnormalities in apparently healthy, physically active individuals. Further research may be warranted to assess long-term cardiovascular outcomes in this population.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 10 years and older
* Consulting for a pre-participation sports medicine evaluation at the Caen University Hospital
* No known history of cardiovascular disease
* Underwent a focused cardiac ultrasound (FCU) of the ascending aorta as part of the consultation
* Consent given for use of anonymized medical data for research purposes

Exclusion Criteria:

* Previous diagnosis of aortic disease or cardiovascular malformation
* Incomplete or non-interpretable FCU images
* Existing cardiology follow-up with echocardiography less than 3 years old
* Refusal to participate or opposition to data use

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes recreational and competitive athletes aged 10 years and older who consulted the Sports Medicine Department at Caen University Hospital for a routine pre-participation cardiovascular evaluation, and who underwent focused cardiac ultrasound of the ascending aorta as part of a standardized screening protocol.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of Ascending Aortic Dilation in Athletes | Baseline
  Proportion of athletes (recreational and competitive) identified with ascending aortic dilation, as determined by focused cardiac ultrasound. Dilation is defined as an aortic diameter ≥ 40 mm and/or a Z-score ≥ 2, according to age-adjusted reference values.

SECONDARY OUTCOMES:
Predictive Factors for Ascending Aortic Dilation | Baseline
  Association between ascending aortic dilation and clinical variables, including age, sex, blood pressure, body mass index, cardiovascular risk factors, and characteristics of physical activity

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Caen Normandie, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided